CLINICAL TRIAL: NCT04552184
Title: A Prospective Single Blinded Randomized SHAM Efficacy Study of Gastric Per Oral Endoscopic Pyloromyotomy (G-POEM) as a Treatment of Gastroparesis
Brief Title: GPOEM Versus SHAM as a Treatement of Gastroparesis
Acronym: GPOEMvsSHAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P2017/334
Record Dates: First submitted 2018-09-05; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPOEM (Active Comparator)
  Interventions: Other: GPOEM
- SHAM (Sham Comparator)
  Interventions: Other: SHAM Procedure

INTERVENTIONS:
Other: GPOEM — gastric per oral endoscopic pyloromyotomy
  Arms: GPOEM
Other: SHAM Procedure — intrapyloric injection of saline solution
  Arms: SHAM

SUMMARY:
Objectives: To evaluate the efficacy of gastric per oral endoscopic pyloromyotomy (G-POEM) in the treatment of gastroparesis.

Endpoints Primary endpoint: Clinical Efficacy Will be assessed by measurements of Gastroparesis Cardinal Symptoms Index (GCSI) score, Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) and the 36-Item Short Form Health Survey (SF-36). Outcome criteria will be measured at baseline, 1 month, 5 months, 7 months and 12 months. These criteria will be the mean total GCSI score, and SF-36 score based on the values recorded with a Likert scale. GES parameters will be the half gastric emptying time and the RPH2.

Secondary endpoint: Safety Safety will be characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants.

In addition, safety assessments will be determined based on physical examination (vital signs) and laboratory tests during scheduled visits. Safety evaluations will also be performed to ensure no subsequent adverse events have occurred and to ensure any adverse events during the trial that are considered on-going are stable or have resolved. Safety will be assessed at 1 month, 5 months, 7 months and 12 months following the intervention.

Other secondary endpoints will be technical success, nutritional status assessed by the measurement of the BMI, pre-albumin and albumin levels and for diabetics the HbA1c. These criteria will be measured at baseline, 1 month, 5 months, 7 months and 12 months.

Overall design This will be a prospective, sham-randomized, monocentric, interventional, efficacy study.

Once baseline eligibility criteria have been met, a first endoscopy under general anesthesia is proposed to the patients. Patients will be randomized blindly in a 1/1 fashion design between the sham arm and the GPOEM arm. At the time of the general anesthesia, a sealed envelope will be opened. Subjects will have a second endoscopy under general anesthesia 6 months later and the sham arm will then beneficiate from a GPOEM procedure and the GPOEM arm a sham procedure. Then, all the patients will be followed for another 6 months.

GCSI score, PAGI-SYM, SF36 will be collected at screening, 1,5,7 and 12 months. GES RPH2, RPH4 and half emptying time will be collected at screening, 5 months and 12 months.

Study procedures

Description procedure in the GPOEM arm:

The intervention will be performed under general anesthesia with tracheal intubation in supine position. GPOEM is performed with the following steps: -i: submucosal injection; -ii: mucosal incision upstream the pylorus followed by submucosal tunneling; -iii: antropyloromyotomy; -iv: closure of the tunnel access.

Description procedure in the SHAM arm:

A diagnostic upper digestive tract endoscopy will be performed under general anesthesia with tracheal intubation in supine position, injection of 1 cc of saline at four quadrants of the pylorus.

Post-operative management Once the patients recovered from anesthesia after the procedure, they were administrated analgesics and anti-emetics as needed and esomeprazole 80 mg daily systematically to protect the mucosal access and tunnel from ulceration. Patients will be kept fasted for the first postoperative day (POD 1). In the absence of adverse events, patients will be allowed to resume liquid oral intake for 1 day, a soft-ground diet for 2 additional days, and finally a normal diet. They will be discharged after POD 1 in the absence of adverse events, with a prescription of esomeprazole 40 mg daily by mouth for 1 month and dietary instructions.

After 6 months, another endoscopy under general anesthesia will be performed with the SHAM and GPOEM arms are interchanged.

After the G-POEM / SHAM procedure, all patients will be rigorously evaluated in the same fashion. They will be assessed clinically before being discharged (POD 1) and then at 1 month and 5 months after the intervention with a clinical examination that included determination of the severity of the symptoms and total GCSI score, PAGI-SYM, SF-36. A GES will be performed at 5 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-64 years;
2. Severe refractory gastroparesis based on the presence of delayed gastric emptying-related symptoms, including nausea, retching, vomiting, abdominal pain, stomach fullness, early satiety, loss of appetite, postprandial fullness, and/or bloating. Dominant symptoms being nausea and vomiting.
3. Severe refractory disease defined by symptoms related to gastroparesis with associated weight loss, failure or recurrence in patients who received available optimal pharmacologic therapies and a Gastroparesis Cardinal Symptoms Index (GCSI) score > 2.3 (calculated as mean of total subscores).
4. Recent (<3 months) upper endoscopy showing no evidence of ulcerative lesions or gastric outlet obstruction
5. Having delayed gastric emptying as defined by a disturbed gastric emptying scintigraphy (GES) study (half emptying time > 100 min).
6. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment, endoscopy, radiography, as well as laboratory investigations.
7. Must be able to understand and be willing to provide written informed consent.

Exclusion Criteria:

1. Achalasia and any other esophageal motility disorders.
2. Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity.
3. Hypertension: uncontrolled hypertension during last 3 month.
4. Severe renal, hepatic, pulmonary disease or cancer.
5. Gastrointestinal stenosis or obstruction.
6. Pregnancy or breastfeeding.
7. Impending gastric surgery 60 days post intervention.
8. Peptic ulcer disease or tumoral lesion at endoscopy.
9. Normal gastric emptying scintigraphy.
10. Presence of coagulation disorders (TP < 50% and/or platelets < 50 G/l), or anesthesiologist exclusion.
11. The chronic use of opioids.
12. Currently participating in other study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 12 months
  Efficacy will be defined by a decrease of a total Gastroparesis Cardinal Symptom Index (GCSI) symptom score of at least 0.75 points from the baseline total score of GCSI
Assessment of Gastrointestinal Disorders Symptom Severity Index | 12 months
  Will be assessed by the significant improvement of the Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM), clinical score from baseline
Quality of life | 12 months
  Quality of Lige will be assessed by the significant improvement of the 36-Item Short Form Health Survey (SF-36), clinical score from baseline

SECONDARY OUTCOMES:
Gastric Emptying Scintigraphy improvement | 12 months
  We will assess significant improvement Gastric Emptying Scintigraphy (GES) parameters from baseline
Safety | 12 months
  Safety will be characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department, Erasme University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided